CLINICAL TRIAL: NCT06018259
Title: Investigations on the Role of Bioactive Lipids in the Control of PBMC Activation and Differentiation.
Brief Title: Bioactive Lipids & PBMC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LIP-PBMC
Record Dates: First submitted 2023-05-04; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental): One blood sample will be taken from healthy volunteers in order to isolate PBMC and to assess the effect of the lipid of interest on them
  Interventions: Procedure: healthy volunteers blood sampling

INTERVENTIONS:
Procedure: healthy volunteers blood sampling — One blood sample will be taken from healthy volunteers in order to isolate PBMC and to assess the effect of the lipid of interest on them PBMC will be activated in vitro (e.g. using LPS or PHA) in the presence or absence of the lipid of interest.

SUMMARY:
The investigators aim at harvesting PBMC from healthy donors to study the effect of the lipids mediators of interest. After isolation from the blood, PBMC will be activated as largely reported in the literature in the presence or absence of the tested lipids. The effect will be assessed by quantifying the expression of inflammatory markers. The expression of the receptors and enzymes potentially regulating the effects of the studied lipids will also be assessed.

DETAILED DESCRIPTION:
Data from the scientific literature support the hypothesis that bioactive lipids play an important role in inflammatory disorders. The levels of these bioactive lipids are altered in several pathophysiological conditions with an inflammatory component. The investigators and others have demonstrated that bioactive lipids affect the inflammatory tone in vivo in murine models as well as in in vitro models. However, confirming the translational value of these data is not easy in clinical studies. PBMC-based experiments are a powerful tool for us to validate our previous observations and will offer translational added value supporting further clinical investigations.

Thus, here the investigators aim at harvesting PBMC from healthy donors and use them to study the effect of the lipid mediators of interest (i.e. those showing interesting properties in our preclinical models). Blood will be collected from healthy volunteers, and PMBC isolated based on their density. After isolation from the blood, PBMC will be activated as largely reported in the literature (e.g. using phytohemagglutinin or lipopolysaccharides) in the presence or absence of the tested lipids. The effect will be assessed by quantifying the expression of inflammatory markers (by RT-qPCR and/or ELISA). The expression of the receptors and enzymes potentially regulating the effects of the studied lipids will be also assessed (by RT-qPCR).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be able to give informed consent to be included in the study.
* no chronic inflammatory disease
* no acute inflammation

Exclusion Criteria:

* Men and women aged less than 18 years
* Pregnant women
* Prior diagnosis of a chronic inflammatory disease (for instance IBD, COPD, lupus, MS, etc. This is not an exhaustive list).
* Recent (<21 days) episode of acute inflammation or immune-altering event (e.g. cold, flu, vaccine, …).
* Chronic or recent use of drugs interfering with the immune / inflammatory response. Examples include (and are not limited to) NSAIDs, corticosteroids, aspirin, mABs, etc.
* Unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Change in PBMC proliferation, differentiation or activation | Throughout the study, an average of 5,5 years
  Expression of inflammatory markers (e.g. cytokines: IL-1, IL-6,...), by RT-qPCR and/or ELISA

SECONDARY OUTCOMES:
Correlation between the expression of enzymes or receptors and the PBMC activation state | Throughout the study, an average of 5,5 years
  Expression of the receptors known to mediate the effects of the lipids studied

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Muccioli, prof, Study Director — Université Catholique de Louvain

IPD SHARING:
Plan to Share IPD: No